CLINICAL TRIAL: NCT00040781
Title: A Phase I Study Of ZD1839 (Iressa TM), An Oral Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor, In Children With Refractory Solid Tumors
Brief Title: Gefitinib in Treating Children With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01874; ADVL0016; U01CA097452 (NIH); CDR0000069406 (Registry Identifier: PDQ (Physician Data Query)); NCT00050739 (obsolete NCT alias)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: interventions — Gefitinib

ARMS (1):
- Treatment (gefitinib) (Experimental): Patients receive oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: gefitinib; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gefitinib — Given orally
  Other Names: Iressa; ZD 1839
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of gefitinib in treating children who have refractory solid tumors. Gefitinib may stop the growth of cancer cells by blocking the enzymes necessary for tumor cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of gefitinib in children with refractory solid tumors.

II. Determine the dose-limiting toxicity of this drug in these patients. III. Determine the pharmacokinetics of this drug in these patients. IV. Determine, preliminarily, the antitumor activity of this drug in these patients.

V. Correlate the pharmacogenetic polymorphisms of this drug with pharmacokinetics and pharmacodynamics in these patients.

OUTLINE: This is a dose-escalation, multicenter study. If myelosuppression is found to be the dose-limiting toxicity, patients are stratified according to prior therapy (more than 2 multiagent chemotherapy regimens or radiotherapy to more than 20% of the bone marrow or stem cell transplantation with or without total body irradiation vs more than 2 single-agent phase I or phase II agents) and extent of disease (bone marrow involvement vs meeting none of the stratum I criteria).

Patients receive oral gefitinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gefitinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 3-45 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor at original diagnosis
* Refractory to conventional therapy and other therapies of higher priority according to the COG Phase I/II priority list or no conventional therapy exists
* No primary CNS tumors or known metastases to the CNS
* Performance status - Karnofsky 50-100% (over 10 years of age)
* Performance status - Lansky 50-100% (10 years of age and under)
* At least 8 weeks
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 50,000/mm^3 (transfusion independent)
* Hemoglobin at least 8.0 g/dL (RBC transfusion allowed)
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 3 times ULN
* Albumin at least 2 g/dL
* Creatinine normal for age
* Glomerular filtration rate at least 70 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* At least 6 months since prior allogeneic stem cell transplantation (SCT)

  * No evidence of active graft-versus-host disease
* At least 1 week since prior biologic agents
* At least 1 week since prior hematopoietic growth factors
* Recovered from prior immunotherapy
* At least 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No concurrent tamoxifen
* At least 2 weeks since prior local palliative (small port) radiotherapy
* At least 6 months since prior craniospinal radiotherapy or radiotherapy to 50% or more of the pelvis (6 weeks for radiotherapy to other substantial amount of bone marrow)
* Recovered from prior radiotherapy
* No concurrent drugs with known corneal toxicity (e.g., chlorpromazine, Amiodarone, or chloroquine)
* No concurrent enzyme-activating anticonvulsants
* No concurrent proton pump inhibitors or H-2 blockers within 4 hours of gefitinib administration

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2002-06; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) based on the incidence of dose-limiting toxicity (DLT) as assessed by the Common Terminology Criteria (CTC) version 2.0 | 28 days
DLT defined as hematologic and non-hematologic toxicities toxicities attributable to drug administration occurring during or immediately subsequent to the first course as assessed by CTC version 2.0 | 28 days
Pharmacokinetics of gefitinib | At baseline, at 1, 2, 4, 6, 8, 12, and 24 hours after administration, at days 21 and 28, and at day 28 of subsequent courses

SECONDARY OUTCOMES:
Antitumor activity of gefitinib according to Response Evaluation Criteria in Solid Tumor (RECIST) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Najat Daw, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States